CLINICAL TRIAL: NCT03339024
Title: Long-term Effects of Intranasal Oxytocin in Alcohol Withdrawal and Dependence: Follow-up of a Randomized Controlled Trial
Brief Title: Intranasal Oxytocin Effects in Alcohol Withdrawal and Dependence; Follow-up Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Lade Addiction Treatment Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016/45; 2015-004463-37 (EudraCT Number)
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Alcoholism; Substance-Related Disorders
Keywords: Oxytocin; Administration, Intranasal; Ethanol; Follow-up Studies
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oxytocin (Experimental): intranasal oxytocin spray Day 1-3: Twice daily intranasal oxytocin spray administered by health personnel.
  Day 3-30:Self-administered intranasal spray as needed, max thrice daily
  Interventions: Drug: intranasal oxytocin spray
- Placebo (Placebo Comparator): intranasal spray without oxytocin Day 1-3: Twice daily intranasal spray without oxytocin, administered by health personnel.
  Day 3-30: Self-administered intranasal spray as needed, max thrice daily
  Interventions: Other: intranasal spray without oxytocin

INTERVENTIONS:
Drug: intranasal oxytocin spray — 6 insufflations (24 IU of oxytocin total) given twice daily, day 1-3. 2 insufflations (8 IU of oxytocin total) as needed, max thrice daily, day 3-30 Day 30 - 12 months: No further oxytocin treatment, i.e. treatment-as-usual.
  Other Names: Syntocinon
  Arms: oxytocin
Other: intranasal spray without oxytocin — 6 insufflations (24 IU of placebo total) given twice daily, day 1-3. 2 insufflations (8 IU of placebo total) as needed, max thrice daily, day 3-30 Day 30 - 12 months: No further oxytocin treatment, i.e. treatment-as-usual.
  Other Names: placebo
  Arms: Placebo

SUMMARY:
This study is an assessment of the long-term effect of oxytocin nasal spray on alcohol withdrawal and dependence in adults admitted for detoxification of alcohol after 60 days and 1 year. It is a follow-up study of a placebo-controlled randomized controlled study where subjects used oxytocin nasal spray during acute withdrawal and the following 4 weeks in an outpatient setting. Half of the participants have received oxytocin nasal spray, the other half placebo nasal spray (NCT02903251). (added March 2019: 24 patients were available for 1-year follow-up)

ELIGIBILITY:
Inclusion Criteria:

* participants in the RCT (NCT02903251) who completed the study

Exclusion Criteria:

* participants in the RCT (NCT02903251) who did not complete the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Alcohol intake | 60 days
  using self-reported alcohol use (days used and alcohol units)
Alcohol intake | 1 year
  using the Timeline Follow-back method and phosphatidylethanol (PEth) blood test

SECONDARY OUTCOMES:
Sleep | 60 days
  self-reported sleeping hours
Sleep | 1 year
  self-reported sleeping hours
Number of rehospitalisations and readmissions to treatment for substance use disorders | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Olav Spigset, MD PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Lade Addiction Treatment Center, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Melby K, Fasmer OB, Henriksen TE, Grawe RW, Aamo TO, Spigset O. Actigraphy assessment of motor activity and sleep in patients with alcohol withdrawal syndrome and the effects of intranasal oxytocin. PLoS One. 2020 Feb 13;15(2):e0228700. doi: 10.1371/journal.pone.0228700. eCollection 2020. PMID 32053696